CLINICAL TRIAL: NCT06557005
Title: Bridges to Primary Care: Transforming Postpartum Primary Care Coordination for People With Chronic Conditions
Brief Title: Facilitated Transitions From Postpartum to Primary Care Coordination for People With Chronic Conditions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Mark Clapp, MD MPH, Physician Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2024P002210; R01HS030245-01 (AHRQ)
Record Dates: First submitted 2024-08-13; First posted 2024-08-16 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Hypertension; Diabetes; Postpartum; Pregnancy; Anxiety; Depression; Obesity
Keywords: Postpartum Care; Primary Care; Care Transitions; Chronic Disease
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Anxiety Disorders; Depression; Obesity; Chronic Disease

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Routine Care (No Intervention): Routine postpartum care
- Facilitated Transition Group (Active Comparator): The intervention is integrated into routine inpatient postpartum care and includes the following components: default PCP visit scheduling, tailored nudge messages to patients, ongoing care recommendations sent to the PCP, and a summary of recommendations after pregnancy given to the patient.
  Interventions: Other: Facilitated Transition to Primary Care

INTERVENTIONS:
Other: Facilitated Transition to Primary Care — The intervention includes default PCP visit scheduling, tailored nudge messages to patients, ongoing care recommendations sent to the PCP, and a summary of recommendations after pregnancy given to the patient.
  Arms: Facilitated Transition Group

SUMMARY:
The lack of postpartum primary care coordination is a missed opportunity to increase primary care engagement and manage chronic conditions early in life, especially for the >30% of pregnant people who have or are at risk for these conditions. This study aims to increase postpartum primary care engagement, quality, and experience by strengthening postpartum transitions to primary care using a behavioral economics-informed, multi-component intervention integrated into usual inpatient postpartum care. Using a randomized controlled trial and repeated outcome assessments through administrative and survey data, this study will generate rigorous, actionable evidence to ensure primary care coordination becomes standard postpartum care practice, potentially catalyzing sustained primary care engagement throughout life.

DETAILED DESCRIPTION:
Over 30% of pregnant people have at least one chronic medical condition, and 20% have certain prenatal conditions (e.g., pregnancy-related hypertension, gestational diabetes) that increase the risk of chronic disease later in life. While patients with these conditions are typically highly engaged in prenatal care, they encounter a "postpartum cliff" in health system support after delivery; many receive no postpartum primary care at all despite having ongoing medical needs. At a time of increased stress, sleep deprivation, and competing demands, they must navigate administrative burdens in accessing primary care, often without scheduling assistance or any formal handoff between their obstetric and primary care clinician (PCP). These burdens may lead to avoided or delayed postpartum primary care, exacerbating health inequities that existed prenatally even for those fortunate enough to have a PCP. Given the many benefits of primary care, this lack of obstetric-to-primary care coordination represents a missed opportunity to increase primary care engagement and manage chronic conditions earlier in life. The primary objective is to increase postpartum primary care engagement, quality, and experience by strengthening obstetric-to-primary care coordination using a behavioral economics-informed intervention. The intervention, integrated into routine inpatient postpartum care, includes default PCP visit scheduling, tailored nudge messages to patients, ongoing care recommendations sent to the PCP, and a summary of recommendations after pregnancy given to the patient. Using a robust randomized controlled trial of 1,320 participants that is built off of the team's pilot study, the proposed study will: (Aim 1) measure the intervention's impact on postpartum primary care visit completion, sustained engagement, and disparities in these outcomes; (Aim 2) measure the intervention's impact on high-value primary care service use; and (Aim 3) measure the intervention's impact on patient experience. The study will generate rigorous, actionable evidence to ensure primary care coordination becomes standard postpartum care practice and will provide insight into postpartum patients' health care experiences. By targeting a vulnerable population at a time of great need and opportunity, postpartum-to-primary care coordination has the potential to catalyze sustained primary care engagement throughout life and improve long-term health.

ELIGIBILITY:
Inclusion Criteria

* Receiving obstetric care at an MGH-affiliated obstetrics practice (except for the MGH HOPE Clinic, which has a unique care model that provides prenatal and postnatal care for individuals with substance use disorder, including the provision of primary care through 2+ years postpartum)
* Pregnant with a live fetus or delivered a live-born neonate ≥24 weeks of gestation, based on the clinical estimate of gestational age
* If postpartum, has a neonate that is currently living at the time of enrollment
* Has one or more of the following conditions listed in the "Problem List," "Medical History," or clinical notes during prenatal, intrapartum, or postpartum encounters in the EHR (or in the case of BMI, the patient's anthropometric measurements):

  * Chronic or essential hypertension
  * Hypertensive disorders related to pregnancy (e.g., pre-eclampsia)
  * Type 1 or 2 diabetes (i.e., pre-existing diabetes)
  * Gestational diabetes
  * Class II Obesity (pre-pregnancy body mass index ≥35 kg/m2; or if pre-pregnancy body mass index is not known, a first trimester BMI of ≥35 kg/m2)
  * Depression or anxiety disorder
* Has a primary care clinician listed in the patient's medical record
* Has access to or agrees to be enrolled in the electronic health record patient portal and consents to be contacted via these modalities
* Able to read/speak English or Spanish language
* Is age ≥18 years old

Exclusion Criteria

• Any individual not meeting all inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1320 (Estimated)
Dates: Start 2025-05-23 (Actual); Primary Completion 2027-05-23 (Estimated); Study Completion 2028-05-23 (Estimated)

PRIMARY OUTCOMES:
Completion of a primary care visit | 155 days after date of delivery
  Observation of a visit with a primary care practitioner (defined as physicians and advanced practice clinicians affiliated with the following medical specialties: internal medicine, family medicine, pediatrics and adolescent medicine, and gynecology).
Receipt of condition-specific recommended health screening and counseling by a primary care practitioner | 155 days after date of delivery
  For individuals with gestational hypertensive disorders, appropriate management is defined as blood pressure screening by a primary care practitioner as documented in the electronic health record.
  For individuals with gestational diabetes, appropriate management is defined as observation of a postpartum glucose screening testing (e.g., GTT, HgbA1c) in the electronic health record.
  For individuals with chronic conditions, appropriate management is defined as receipt of both condition-specific screening (mood, weight, blood pressure and/or diabetes screening) and receipt of counseling, discussion of a management, and/or referral for or acknowledgment of subspecialist management for that condition by a primary care practitioner as documented in the electronic health record. "
Self-report of having a known, reliable primary care practitioner | 155 days after date of delivery
  The outcome is the Self-report of having a known, reliable primary care practitioner (doctor, nurse practitioner, or physician's assistant).
Self-report of mental health | 155 days after date of delivery
  Edinburgh Perinatal Depression Scale will be administered and the total EPDS score compared.

SECONDARY OUTCOMES:
Completion of an annual exam with a primary care practitioner | 155 days after date of delivery
  Observation of an annual exam or health care maintenance visit with a primary care practitioner (defined as physicians and advanced practice clinicians affiliated with the following medical specialties: internal medicine, family medicine, pediatrics and adolescent medicine, and gynecology).
Self-report of completion of a primary care visit | 155 days after date of delivery
  Self-report of a visit with a primary care practitioner (defined as physicians and advanced practice clinicians affiliated with the following medical specialties: internal medicine, family medicine, pediatrics and adolescent medicine, and gynecology) for any reason.
Self-report of an annual exam with a primary care practitioner | 155 days after date of delivery
  Self-report of an annual exam or health care maintenance visit with a primary care practitioner (defined as physicians and advanced practice clinicians affiliated with the following medical specialties: internal medicine, family medicine, pediatrics and adolescent medicine, and gynecology).
Completion of a primary care visit | 365 days after date of delivery
  Observation of a visit with a primary care practitioner for any reason.
Self-report of completion of a primary care visit | 365 days after date of delivery
  Self-report of a visit with a primary care practitioner (defined as physicians and advanced practice clinicians affiliated with the following medical specialties: internal medicine, family medicine, pediatrics and adolescent medicine, and gynecology) for any reason.
Completion of an annual exam with a primary care practitioner | 365 days after date of delivery
  Observation of an annual exam or health care maintenance visit with a primary care practitioner (defined as physicians and advanced practice clinicians affiliated with the following medical specialties: internal medicine, family medicine, pediatrics and adolescent medicine, and gynecology).
Self-report of an annual exam with a primary care practitioner | 365 days after date of delivery
  Self-report of an annual exam or health care maintenance visit with a primary care practitioner (defined as physicians and advanced practice clinicians affiliated with the following medical specialties: internal medicine, family medicine, pediatrics and adolescent medicine, and gynecology).
Repeated primary care practitioner engagement | 365 days after date of delivery
  Observation of two or more primary care practitioner visits for any reason.
Self-report of repeated primary care practitioner engagement | 365 days after date of delivery
  Self-report of two or more primary care practitioner visits for any reason.
Extent of primary care practitioner engagement | 365 days after date of delivery
  Number of primary care practitioner visits for any reason.
Self-report of extent of primary care practitioner engagement | 365 days after date of delivery
  Self-report of the number of primary care practitioner visits for any reason.
Completion of a primary care visit | 548 days after date of delivery
  Observation of a visit with a primary care practitioner for any reason.
Completion of an annual exam with a primary care practitioner | 548 days after date of delivery
  Observation of an annual exam or health care maintenance visit with a primary care practitioner.
Repeated primary care practitioner engagement | 548 days after date of delivery
  Observation of two or more primary care practitioner visits for any reason.
Extent of primary care practitioner engagement | 548 days after date of delivery
  Number of primary care practitioner visits for any reason.
Self-report of receipt of condition-specific recommended health screening and counseling by a primary care practitioner | 155 days after date of delivery
  For individuals with gestational hypertensive disorders, appropriate management is defined as blood pressure screening by a primary care practitioner as reported by the participant.
  For individuals with gestational diabetes, appropriate management is defined as observation of a postpartum glucose screening testing (e.g., GTT, HgbA1c) as reported by the participant.
  For individuals with chronic conditions, appropriate management is defined as receipt of both condition-specific screening (mood, weight, blood pressure and/or diabetes screening) and receipt of counseling, discussion of a management, and/or referral for or acknowledgment of subspecialist management for that condition by a primary care practitioner as reported by the participant.
Receipt of recommended screening and counseling for chronic condition by primary care practitioner | 155 days after date of delivery
  For individuals with chronic conditions, appropriate management is defined as receipt of both condition-specific screening (mood, weight, blood pressure and/or diabetes screening) and receipt of counseling, discussion of a management, and/or referral for or acknowledgment of subspecialist management for that condition by a primary care practitioner as documented in the electronic health record.
Receipt of recommended screening for gestational condition by primary care practitioner | 155 days after date of delivery
  For individuals with gestational hypertensive disorders, appropriate management is defined as blood pressure screening by a primary care practitioner as documented in the electronic health record.
  For individuals with gestational diabetes, appropriate management is defined as observation of a postpartum glucose screening testing (e.g., GTT, HgbA1c) in the electronic health record."
Receipt of recommended screening and counseling for chronic condition by primary care practitioner | 365 days after date of delivery
  For individuals with chronic conditions, appropriate management is defined as receipt of both condition-specific screening (mood, weight, blood pressure and/or diabetes screening) and receipt of counseling, discussion of a management, and/or referral for or acknowledgment of subspecialist management for that condition by a primary care practitioner as documented in the electronic health record.
Receipt of recommended screening for gestational condition by primary care practitioner | 365 days after date of delivery
  For individuals with gestational hypertensive disorders, appropriate management is defined as blood pressure screening by a primary care practitioner as documented in the electronic health record.
  For individuals with gestational diabetes, appropriate management is defined as observation of a postpartum glucose screening testing (e.g., GTT, HgbA1c) in the electronic health record.
Receipt of recommended screening and counseling for chronic condition by primary care practitioner | 548 days after date of delivery
  For individuals with chronic conditions, appropriate management is defined as receipt of both condition-specific screening (mood, weight, blood pressure and/or diabetes screening) and receipt of counseling, discussion of a management, and/or referral for or acknowledgment of subspecialist management for that condition by a primary care practitioner as documented in the electronic health record.
Receipt of recommended screening for gestational condition by primary care practitioner | 548 days after date of delivery
  For individuals with gestational hypertensive disorders, appropriate management is defined as blood pressure screening by a primary care practitioner as documented in the electronic health record.
  For individuals with gestational diabetes, appropriate management is defined as observation of a postpartum glucose screening testing (e.g., GTT, HgbA1c) in the electronic health record.
Self-report of receipt of recommended screening and counseling for chronic condition by primary care practitioner | 365 days after date of delivery
  For individuals with chronic conditions, appropriate management is defined as receipt of both condition-specific screening (mood, weight, blood pressure and/or diabetes screening) and receipt of counseling, discussion of a management, and/or referral for or acknowledgment of subspecialist management for that condition by a primary care practitioner as reported by the participant.
Self-report of receipt of recommended screening for gestational condition by primary care practitioner | 365 days after date of delivery
  For individuals with gestational hypertensive disorders, appropriate management is defined as blood pressure screening by a primary care practitioner as reported by the participant.
  For individuals with gestational diabetes, appropriate management is defined as observation of a postpartum glucose screening testing (e.g., GTT, HgbA1c) as reported by the participant. "
Self-report of having a known, reliable primary care practitioner | 365 days after date of delivery
  Participant report of having a known, reliable primary care practitioner (doctor, nurse practitioner, or physician's assistant).
Urgent or emergent care use | 155 days after date of delivery
  Emergency department or urgent care visit for any reason as documented in the electronic health record.
Self-report of urgent or emergent care use | 155 days after date of delivery
  Emergency department or urgent care visit for any reason as documented as reported by the participant.
Urgent or emergent care use | 365 days after date of delivery
  Emergency department or urgent care visit for any reason as documented in the electronic health record.
Self-report of urgent or emergent care use | 365 days after date of delivery
  Emergency department or urgent care visit for any reason as reported by the participant.
Self-report of mental health | 365 days after date of delivery
  Edinburgh Perinatal Depression Scale score as reported by the participant.
Urgent or emergent care use | 584 days after date of delivery
  Emergency department or urgent care visit for any reason as documented in the electronic health record.
Interpregnancy interval | 365 days after date of delivery
  Defined as the time (in days) from date of delivery until subsequent date of conception.
Interpregnancy interval | 584 days after date of delivery
  Defined as the time (in days) from date of delivery until subsequent date of conception.
Prescription or documentation of medication use for the treatment of a pre-existing or newly diagnosed mood or anxiety disorder | 155 days
  Observation of a prescription for or provider documentation noting the use of a medication for the treatment of a pre-existing or newly diagnosed mood or anxiety disorder in the electronic health record.
Prescription or documentation of medication use for the treatment of a pre-existing or newly diagnosed mood or anxiety disorder | 365 days
  Observation of a prescription for or provider documentation noting the use of a medication for the treatment of a pre-existing or newly diagnosed mood or anxiety disorder in the electronic health record.
Prescription or documentation of medication use for the treatment of a pre-existing or newly diagnosed mood or anxiety disorder | 584 days
  Observation of a prescription for or provider documentation noting the use of a medication for the treatment of a pre-existing or newly diagnosed mood or anxiety disorder in the electronic health record.
Contraception use | 155 days
  The use of any form of contraception as documented in the electronic health record
Contraception use | 365 days
  The use of any form of contraception as documented in the electronic health record
Contraception use | 584 days
  The use of any form of contraception as documented in the electronic health record
Self-report of contraception | 155 days
  Self-report of using contraception or discussing family planning/contraception
Self-report of contraception | 365 days
  Self-report of using contraception or discussing family planning/contraception

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Clapp, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sets generated for this analysis will be preserved and shared publicly after planned primary and secondary analyses are completed by the research team or at the end of the award, whichever occurs last. Data will be preserved for at least 5 years after public posting to ensure outside investigators can access and use this information for related research.
  Study metadata, code, and a deidentified data set that includes all collected trial data will be publicly available, without restricted access, on the Harvard Dataverse Repository.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data and materials will be available after planned primary and secondary analyses are completed by the research team or at the end of the award, whichever occurs last (expected 08/2029). Data will be available and accessible for at least 5 years after posting.
Access Criteria: Study metadata, code, and a deidentified data set that includes all collected trial data will be publicly available, without restricted access, on the Harvard Dataverse Repository
URL: https://dataverse.harvard.edu/